CLINICAL TRIAL: NCT04535921
Title: Fear of Cancer Recurrence in Malignant Diseases of the Genitourinary Tract
Brief Title: Fear of Cancer Recurrence in Genitourinary Cancer
Status: Completed | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Yannic Volz, Assistant doctor, Ludwig-Maximilians - University of Munich
Other Study IDs: FCR2020
Record Dates: First submitted 2020-08-27; First posted 2020-09-02 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Fear of Cancer Recurrence; Prostate Cancer; Renal Cell Cancer; Urothelial Carcinoma; Testicle Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Carcinoma, Renal Cell; Carcinoma, Transitional Cell; Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Prostatectomy: FCR7 questionnaire pre and postoperative
  Interventions: Other: FCR7 questionnaire
- Cystectomy: FCR7 questionnaire pre and postoperative, 6 months follow
  Interventions: Other: FCR7 questionnaire
- Nephrectomy: FCR7 questionnaire pre and postoperative
  Interventions: Other: FCR7 questionnaire
- Orchidectomy: FCR7 questionnaire pre and postoperative
  Interventions: Other: FCR7 questionnaire

INTERVENTIONS:
Other: FCR7 questionnaire — A 7 item questionnaire about fear of cancer recurrence

SUMMARY:
To perform an analysis of independent predictors of fear of cancer recurrence in patients with malignant genitourinary diseases and their impact on quality of life and survival

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed diagnosis of either prostate, urothelial cell, testicular or renal cell cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed genitourinary malignant disease undergoing curative surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in fear of cancer recurrence pre- and postoperatively | 7 to 10 days after initial surgery
  Changes in the FCR7 score pre- and postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Ludwig-Maximilian-Universität, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No